CLINICAL TRIAL: NCT01890473
Title: Phase Ib, Multicenter, Randomized, Open-Label, Parallel-Group Study to Characterize the Pharmacokinetics of a Single Dose of Abatacept 125 mg Administered Subcutaneously Using the BD Physioject™ Autoinjector or the UltraSafe Passive Needle Guard Prefilled Syringe
Brief Title: Study to Characterize the Pharmacokinetics of a Single Dose of SC Abatacept 125 mg Using the BD Autoinjector or the Prefilled Syringe
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IM101-366
Record Dates: First submitted 2013-06-27; First posted 2013-07-01 (Estimated); Results first posted 2015-11-26 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2015-10

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Abatacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1: Abatacept (autoinjector) (Experimental): Abatacept 125 mg/syringe subcutaneously through autoinjector, one dose in 71 days
  Interventions: Drug: Abatacept
- Arm 2: Abatacept (prefilled syringe) (Experimental): Abatacept 125 mg/syringe subcutaneously with prefilled syringe, one dose in 71 days
  Interventions: Drug: Abatacept

INTERVENTIONS:
Drug: Abatacept
  Other Names: Orencia; BMS-188667

SUMMARY:
The primary purpose of the protocol is to describe the pharmacokinetics of a single dose of Abatacept 125 mg in Rheumatoid Arthritis patients delivered via the autoinjector device or the approved prefilled syringe.

DETAILED DESCRIPTION:
SC=Subcutaneous

ELIGIBILITY:
Key Inclusion Criteria:

* Subjects ≥18 years of age
* Diagnosis of Rheumatoid Arthritis confirmed by participant's physician
* Disease activity under control

Key Exclusion Criteria:

* Change in disease-modifying antirheumatic drug (DMARD) therapy within 3 months of enrollment
* Exposure to investigational drug within 4 weeks or 5 half lives whichever is longer
* Current or prior use of Rituximab ≤6 months
* Current or prior use of the following within 4 weeks or 5 half lives whichever is longer: biologic DMARDS, Tofacitinib, Cyclophosphamide, Mycophenolate Mofetil & d-Penicillamine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 356 (Actual)
Dates: Start 2013-07; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (22):
- United States (13):
  - Rheumatology Associates Of North Alabama, P.C., Huntsville, Alabama
  - Immunoe Int'L Research Ctrs, Centennial, Colorado
  - Covance Cru Inc, Daytona Beach, Florida
  - Heartland Research Associates, Llc, Wichita, Kansas
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - Physician Research Collaboration, Llc, Lincoln, Nebraska
  - Djl Research, Pllc, Charlotte, North Carolina
  - Wake Research Associates, Raleigh, North Carolina
  - Pmg Research Of Salisbury, Salisbury, North Carolina
  - Pmg Research Of Wilmington Llc, Wilmington, North Carolina
  - Community Research, Cincinnati, Ohio
  - Altoona Center For Clinical Research, Duncansville, Pennsylvania
  - Covance Clinical Research Unit Inc., Dallas, Texas
- Argentina (4):
  - Local Institution, San Fernando, Buenos Aires
  - Local Institution, Córdoba, Córdoba Province
  - Local Institution, Rosario, Santa Fe Province
  - Local Institution, San Miguel de Tucumán, Tucumán Province
- Local Institution, Yucatán, Yucatán, Mexico
- Local Institution, Lima, Lima Province, Peru
- South Africa (3):
  - Local Institution, Port Elizabeth, Eastern Cape
  - Local Institution, Pretoria, Gauteng
  - Local Institution, George, Western Cape

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 356 participants enrolled and 224 randomized. 132 not randomized and reasons for non-randomization: 106 no longer met study criteria, 15 other, 9 withdrew consent, and 2 lost to follow-up.
Groups:
- 125 mg Abatacept Via Autoinjector: A single dose of 125 mg abatacept was administered subcutaneously (SC) via an autoinjector.
- 125 mg Abatacept Via Prefilled Syringe: A single dose of 125 mg abatacept was administered SC via a Prefilled Syringe (PFS).
Period: Overall Study
Arm/Group | 125 mg Abatacept Via Autoinjector | 125 mg Abatacept Via Prefilled Syringe
Started | 111 | 113
Completed | 109 | 113
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Poor/non-compliance | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants were summarized.
Groups:
- Total: Total of all reporting groups
Arm/Group | 125 mg Abatacept Via Autoinjector | 125 mg Abatacept Via Prefilled Syringe | Total
Number analyzed (Participants) | 111 | 113 | 224
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.0 (13.34) | 56.8 (12.36) | 54.9 (12.97)
Age, Customized [Number; unit: participants]
  Less than (<) 65 | 90 | 75 | 165
  Greater than, equal to (>=) 65 | 21 | 38 | 59
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90 | 87 | 177
  Male | 21 | 26 | 47

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Geometric Mean of Maximum Observed Serum Concentration (Cmax) of a Single Dose of Subcutaneous (SC) Abatacept - PK-Evaluable Analysis Population
Description: Serum concentrations of abatacept were analyzed using a validated enzyme-linked immunosorbent assay (ELISA). Cmax was measured in micrograms per milliliter (μg/mL). Blood samples for pharmacokinetic (PK) parameters were collected at Day 1 pre-dose at 0 hour (h), 1, 2, and 8 h post dose, and on subsequent Days, 2 (24 h post dose), 3 (48 h), 5 (96 h), 8 (168 h), 15 (336 h), 29 (672 h) , 43 (1008 h), 57 (1344 h) and 71 (1680 h) following the single administration of abatacept SC.
Time Frame: Day 1 to Day 71
Population: PK-evaluable analysis population: All randomized and treated participants with adequately evaluable PK parameters were summarized.
Measure: Geometric Mean (90% Confidence Interval); unit: μg/mL
Arm/Group | 125 mg Abatacept Via Autoinjector | 125 mg Abatacept Via Prefilled Syringe
Number analyzed (Participants) | 105 | 111
μg/mL | 11.5 [10.6 to 12.4] | 12.6 [11.7 to 13.6]
Statistical Analysis 1: Comparison: 125 mg Abatacept Via Autoinjector vs 125 mg Abatacept Via Prefilled Syringe; The PK comparability of the two devices was assessed via a linear model for each key PK parameter in log scale (using log (Cmax) without a formal test; Test type: Superiority or Other; ratio of geometric mean = 0.908, 90% CI 2-sided [0.815 to 1.01]

2. Primary Outcome: Adjusted Geometric Mean of Area Under the Serum Concentration-time Curve (AUC) From Zero to the Last Time of the Last Quantifiable Concentration (0-T) of a Single Dose of SC Abatacept - PK-Evaluable Analysis Population
Description: Serum concentrations of abatacept were analyzed using ELISA. AUC (0-T) was measured in μg*h/mL. Blood samples were collected at Day 1 pre-dose at 0 h, 1, 2, and 8 h post dose, and on subsequent Days, 2 (24 h post dose), 3 (48 h), 5 (96 h), 8 (168 h), 15 (336 h), 29 (672 h) , 43 (1008 h), 57 (1344 h) and 71 (1680 h) following the single administration of abatacept SC.
Time Frame: Day 1 to Day 71
Population: as for outcome 1
Measure: Geometric Mean (90% Confidence Interval); unit: μg*h/mL
Groups:
- 125 mg Abatacept Via Autoinjector: A single dose of 125 mg abatacept was administered SC via an autoinjector.
- 125 mg Abatacept Via Prefilled Syringe: A single dose of 125 mg abatacept was administered SC via a Prefilled Syringe.
Arm/Group | 125 mg Abatacept Via Autoinjector | 125 mg Abatacept Via Prefilled Syringe
Number analyzed (Participants) | 105 | 111
μg*h/mL | 4991 [4613 to 5400] | 5304 [4913 to 5727]
Statistical Analysis 1: Comparison: 125 mg Abatacept Via Autoinjector vs 125 mg Abatacept Via Prefilled Syringe; The PK comparability of the two devices was assessed via a linear model for each key PK parameter in log scale, using log (AUC (0-T) without a formal test; Test type: Superiority or Other; ratio of geometric mean = 0.941, 90% CI 2-sided [0.843 to 1.05]

3. Primary Outcome: Adjusted Geometric Mean of Area Under the Serum Concentration-time Curve From Time Zero to Extrapolated to Infinity, AUC (INF), of a Single Dose of SC Abatacept - PK-Evaluable Analysis Population
Description: Serum concentrations of abatacept were analyzed using ELISA. Blood samples were collected at Day 1 pre-dose at 0 hour (h), 1, 2, and 8 h post dose, and on subsequent Days, 2 (24 h post dose), 3 (48 h), 5 (96 h), 8 (168 h), 15 (336 h), 29 (672 h) , 43 (1008 h), 57 (1344 h) and 71 (1680 h) following the single administration of abatacept SC. AUC (INF) was measured in μg*h/mL
Time Frame: Day 1 to Day 71
Population: as for outcome 1
Measure: Geometric Mean (90% Confidence Interval); unit: μg*h/mL
Arm/Group | 125 mg Abatacept Via Autoinjector | 125 mg Abatacept Via Prefilled Syringe
Number analyzed (Participants) | 104 | 111
μg*h/mL | 5308 [4957 to 5684] | 5437 [5089 to 5810]
Statistical Analysis 1: Comparison: 125 mg Abatacept Via Autoinjector vs 125 mg Abatacept Via Prefilled Syringe; The PK comparability of the two devices was assessed via a linear model for each key PK parameter in log scale, using log AUC(INF) without a formal test; Test type: Superiority or Other; ratio of geometric mean = 0.976, 90% CI 2-sided [0.888 to 1.07]

4. Secondary Outcome: Median of Time to Reach Cmax in Serum (Tmax) of a Single Dose of SC Abatacept - PK-Evaluable Analysis Population
Description: Serum concentrations of abatacept were analyzed using ELISA. Blood samples were collected at Day 1 pre-dose at 0 h, 1, 2, and 8 h post dose, and on subsequent Days, 2 (24 h post dose), 3 (48 h), 5 (96 h), 8 (168 h), 15 (336 h), 29 (672 h) , 43 (1008 h), 57 (1344 h) and 71 (1680 h) following the single administration of abatacept SC. Tmax was measured in hours (h).
Time Frame: Day 1 to Day 71
Population: as for outcome 1
Measure: Median (Full Range); unit: h
Arm/Group | 125 mg Abatacept Via Autoinjector | 125 mg Abatacept Via Prefilled Syringe
Number analyzed (Participants) | 105 | 111
h | 96.0 [24 to 337] | 96.0 [24 to 336]

5. Secondary Outcome: Mean of Terminal Phase Elimination Half-life in Serum (T-HALF) of a Single Dose of SC Abatacept - PK-Evaluable Analysis Population
Description: Serum concentrations of abatacept were analyzed using ELISA. Blood samples were collected at Day 1 pre-dose at 0 h, 1, 2, and 8 h post dose, and on subsequent Days, 2 (24 h post dose), 3 (48 h), 5 (96 h), 8 (168 h), 15 (336 h), 29 (672 h) , 43 (1008 h), 57 (1344 h) and 71 (1680 h) following the single administration of abatacept SC. T-HALF was measured in hours (h).
Time Frame: Day 1 to Day 71
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h
Arm/Group | 125 mg Abatacept Via Autoinjector | 125 mg Abatacept Via Prefilled Syringe
Number analyzed (Participants) | 104 | 111
h | 285 (89.54) | 302 (99.82)

6. Secondary Outcome: Geometric Mean of Total Body Clearance (CL/F) of a Single Dose of SC Abatacept - PK-Evaluable Analysis Population
Description: Serum concentrations of abatacept were analyzed using ELISA. Blood samples were collected at Day 1 pre-dose at 0 h, 1, 2, and 8 h post dose, and on subsequent Days, 2 (24 h post dose), 3 (48 h), 5 (96 h), 8 (168 h), 15 (336 h), 29 (672 h) , 43 (1008 h), 57 (1344 h) and 71 (1680 h) following the single administration of abatacept SC. CL/F was measured in milliliters per hour per kilogram body weight (mL/h/kg).
Time Frame: Day 1 to Day 71
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/h/kg
Arm/Group | 125 mg Abatacept Via Autoinjector | 125 mg Abatacept Via Prefilled Syringe
Number analyzed (Participants) | 104 | 111
mL/h/kg | 0.31 (52) | 0.30 (62)

7. Secondary Outcome: Geometric Mean of Volume of Distribution (V/F) of a Single Dose of Subcutaneous (SC) Abatacept - PK-Evaluable Analysis Population
Description: Serum concentrations of abatacept were analyzed using ELISA. Blood samples were collected at Day 1 pre-dose at 0 h, 1, 2, and 8 h post dose, and on subsequent Days, 2 (24 h post dose), 3 (48 h), 5 (96 h), 8 (168 h), 15 (336 h), 29 (672 h) , 43 (1008 h), 57 (1344 h) and 71 (1680 h) following the single administration of abatacept SC. V/F was measured in liters per kilogram body weight (L/kg)
Time Frame: Day 1 to Day 71
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/kg
Arm/Group | 125 mg Abatacept Via Autoinjector | 125 mg Abatacept Via Prefilled Syringe
Number analyzed (Participants) | 104 | 111
L/kg | 0.12 (43) | 0.12 (62)

8. Secondary Outcome: Number of Participants Who Had Serious Adverse Events (SAEs), Adverse Events (AEs) That Led to Discontinuation, or Who Died
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Treatment-related=having certain, probable, possible, or missing relationship to study drug. Includes data Day 1 up to 76 days (71 days + 5 day window) post the single dose of study drug.
Time Frame: Day 1 to 76 days post single dose
Population: All treated participants were included in safety analysis.
Measure: Number; unit: participants
Arm/Group | 125 mg Abatacept Via Autoinjector | 125 mg Abatacept Via Prefilled Syringe
Number analyzed (Participants) | 111 | 113
participants
  Death | 0 | 0
  SAE | 0 | 1
  Related SAEs | 0 | 0
  Discontinued due to AE | 0 | 0

9. Secondary Outcome: Number of Participants With Adverse Events of Special Interest
Description: Prospectively identified events of special interest which were a subset of all AEs, and were either SAEs or non-serious AEs, included the following categories: Infections, Autoimmune Disorders, Malignancy, local site reactions, any AE occurring within 24 hours of SC injection. AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization.
Time Frame: Day 1 to 76 days post single dose
Population: All treated participants were included in safety analysis.
Measure: Number; unit: participants
Arm/Group | 125 mg Abatacept Via Autoinjector | 125 mg Abatacept Via Prefilled Syringe
Number analyzed (Participants) | 111 | 113
participants
  Infections | 19 | 17
  Autoimmune Disorders | 0 | 0
  Malignancy | 0 | 0
  Local site reactions | 1 | 3
  AEs within 24 hours of SC injection | 10 | 7

10. Secondary Outcome: Number of Participants With a Positive Immunogenicity Response Relative to Baseline
Description: Blood samples were screened at baseline, Day 57 and Day 71 for the presence of drug-specific antibodies using Electrochemiluminescence (ECL). A positive immunogenicity response relative to baseline for Anti-Cytotoxic T Lymphocyte Antigen 4-T Cell (CTLA4) and 'possibly immunoglobulin (Ig)', and 'Ig and/or Junction Region', respectively, was defined as: A missing baseline immunogenicity measurement and a positive analytical laboratory reported immunogenicity response post-baseline; A negative baseline immunogenicity response and a positive analytical laboratory reported immunogenicity response post-baseline; A positive baseline immunogenicity response and a positive analytical laboratory reported immunogenicity response post-baseline that has a titer value strictly greater than the baseline titer value. Baseline=Pre-dose value.
Time Frame: Day 57, Day 71
Population: All treated participants with at least one post baseline immunogenicity result reported were included in the immunogenicity analysis. n=number of participants evaluated at the specific time point.
Measure: Number; unit: participants
Arm/Group | 125 mg Abatacept Via Autoinjector | 125 mg Abatacept Via Prefilled Syringe
Number analyzed (Participants) | 109 | 113
participants
  Day 57 CTLA4, possibly Ig (n=109,111) | 10 | 13
  Day 57 Ig and/or junction (n=109,111) | 4 | 5
  Day 71 CTLA4, possibly Ig (n=105,112) | 23 | 22
  Day 71 Ig and/or junction (n=105,112) | 1 | 5
  Overall CTLA4, possibly Ig (n=109,113) | 24 | 24
  Overall Ig and/or junction (n=109,113) | 4 | 8

11. Secondary Outcome: Number of Participants With Blood Hematology, Chemistry Laboratory Values and Urinalysis Laboratory Values Meeting the Marked Abnormality Criteria
Description: Marked abnormality criteria: lower limit of normal (LLN); upper limit of normal (ULN); pretreatment (preRX); cells per microliter (cµ/L); milligram per deciliter (mg/dL); milliequivalent (mEq): Hematology: leukocytes (*10^3 c/µL): <0.75*LLN or >1.25*ULN, or if preRX <LLN, use <0.8*preRX or >ULN, or if preRX>ULN, use >1.2*preRX or <LLN; eosinophils (*10^3 cµ/L): if value >0.750*10^3 c/µL; lymphocytes (*10^3 cµ/L): if value <0.750*10^3 c/µL or if value >7.50*10^3 c/µL. Chemistry: blood urea nitrogen (mg/dL): >2*preRX; creatinine (mg/dL): >1.5*preRX; potassium (mEq/L): <0.9*LLN or >1.1*ULN, or if preRX<LLN, use <0.9*preRX or >ULN, or if preRX>ULN, use 1.1*preRX or <LLN; glucose (mg/dL): <65 mg/dL (low) or >220 mg/dL (high). Urine Blood, urine red blood cell (RBC), urine white blood cell (WBC): if missing PreRX use >= 2, or if Value >= 4, or if preRX = 0 or 0.5 then use >= 2, or if preRX = 1 then use >= 3, or if preRX = 2 or 3 then use >= 4.
Time Frame: Day 1 to 76 days post last dose
Population: All treated participants with laboratory values were included in the safety analysis. n=number of participants evaluated.
Measure: Number; unit: participants
Arm/Group | 125 mg Abatacept Via Autoinjector | 125 mg Abatacept Via Prefilled Syringe
Number analyzed (Participants) | 111 | 113
participants
  Leukocytes High (n=109, 110) | 1 | 0
  Leukocytes Low (n=109, 110) | 0 | 1
  Eosinophils High (n=107,107) | 1 | 0
  Lymphocytes Low (n=107,107) | 2 | 5
  Blood Urea Nitrogen High (n=109,111) | 1 | 0
  Creatinine High (n=109,111) | 2 | 0
  Potassium Low (n=109,111) | 0 | 1
  Glucose High (n=109,110) | 2 | 0
  Glucose Low (n=109,110) | 3 | 3
  Urine Blood High (n=104,107) | 7 | 1
  Urine RBC High (n=28, 26) | 5 | 2
  Urine WBC High (n=35, 33) | 11 | 13

ADVERSE EVENTS:
Groups:
- 125 mg Abatacept Via Prefilled Syringe: A single dose of 125 mg abatacept was administered SC via a PFS.
Arm/Group | 125 mg Abatacept Via Autoinjector | 125 mg Abatacept Via Prefilled Syringe
Serious Adverse Events (participants affected / at risk) | 0/111 | 1/113
Other Adverse Events (participants affected / at risk) | 0/111 | 0/113
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 125 mg Abatacept Via Autoinjector (N=111) | 125 mg Abatacept Via Prefilled Syringe (N=113)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.